CLINICAL TRIAL: NCT05643443
Title: Effect of Gradually Increasing Force Magnitude on the Rate of Canine Retraction: A Split Mouth Randomized Controlled Trial
Brief Title: Effect of Gradually Increasing Force Magnitude on the Rate of Canine Retraction Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shady Abd ElSalam Rizk ElEsh, Principal Investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ORTH 3-3-3-3
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Canine Retraction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control Group
- Active Group (Experimental): Active Group
  Interventions: Other: Gradual increase of force

INTERVENTIONS:
Other: Gradual increase of force — steady force
  Other Names: 150 gm
  Arms: Active Group

SUMMARY:
Therefore the aim of the current randomized controlled clinical trial is to investigate the effect of gradually increasing force magnitude versus constant force magnitude on the rate of tooth movement in a canine retraction model, furthermore investigate the effect of the two force systems on the ratio of cytokines and the pain experienced by the patient.

Research question:

In adult orthodontic patients requiring bilateral maxillary canines retraction, will gradually increasing force magnitudes accelerate the rate of canine retraction in the experimental side when compared to the control side?

DETAILED DESCRIPTION:
A. -Patient preparation:

1. After patient selection, routine orthodontic records will be collected (study models, panoramic, lateral cephalometric radiographs, and intra-oral and extra-oral photographs).
2. The orthodontic treatment: All subjects will receive a Straight Wire Appliance (SWA); Roth prescription slot 0.022 × 0.028 inch. The brackets will be bonded to the tooth surface using orthodontic light cured composite resin. Ready-made molar bands with 2 buccal tubes (main and auxiliary)1 will be selected, fitted, and cemented on the upper first molars using glass ionomer cement. The arch wire sequence in the initial levelling and alignment stage will be tailored according to the severity of crowding of each case.
3. Just before canine retraction, alginate impressions will be made for the maxillary arch, CGF sample will be taken as described later in the same section, stainless steel arch wire 0.017 x 0.025 mil will be inserted.

B. Canine Retraction:

1. The active group (gradually increasing force magnitude) will be randomly assigned to either the patients' left or right sides only (split mouth design).
2. At the start of canine retraction, Nickel-titanium closed-coil springs applying 50 g and 150 g measured using Correx tension gauge will be used in the active side and control sides respectively on each side, stretched bilaterally from the hook on the first molar band to the hook of canine brackets(19).
3. Activation will be done every 4 weeks.
4. The impressions will be poured with dental stone within 15 minutes to ensure its accuracy.
5. Visual analogue scale (VAS) will be explained to the patient and used to measure pain intensity in the postoperative period: immediately after the commencement of canine retraction and at each visit. The patient is asked to make three pain ratings each time to take an average. (one day, second day and one week after)

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females with an age ranging between 16-30 years (Adult patients since cooperation increases with age) (17).
2. Malocclusion that requires extraction of the maxillary first premolars and canines retraction with moderate anchorage.
3. Full permanent dentition with exception of the third molars.
4. Good oral hygiene and periodontal condition (Probing depth< 4 mm in all teeth), since the periodontal condition affects the amount and type of tooth movement.
5. Absence of untreated caries which may worsen during the study time.

Exclusion Criteria:

1. Medically compromised patients.
2. Patients suffering from any congenital or hereditary diseases.
3. Smoking or any systemic diseases.
4. Chronic use of any medications including antibiotics, phenytoin, cyclosporine, anti-inflammatory drugs, systemic corticosteroids, and calcium channel blockers. All the above factors affect the rate of tooth movement

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | 4 months
  mm/time
change on the Cytokine levels in the gingival crevicular fluid | 3 months
  ratio

SECONDARY OUTCOMES:
The effect of gradually increasing force magnitude on Pain | 4 months
  numeric Pain scale ( 0 as no Pain - 10 As maximum Pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Salah Fayed, Professor, Study Chair — Cairo University, Faculty of Dentistry
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No